CLINICAL TRIAL: NCT05979012
Title: Jazz Music and Mindfulness for Chronic Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Sean D Young, Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3454
Record Dates: First submitted 2023-07-28; First posted 2023-08-07 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Jazz Only (Active Comparator): Jazz Group 1: Participants in this group will watch an introduction to jazz appreciation video prior to the 4-week intervention.
  Interventions: Behavioral: Listening to Jazz
- MIndfullness and Jazz (Experimental): Jazz Group 2 (Mindful Jazz) Group: Participants in this group will watch an introduction to jazz appreciation and mindfulness training video, including the use of jazz for pain tolerance prior to the 4-week intervention.
  Interventions: Behavioral: MIndfulness Listening to Jazz
- Waitlist (No Intervention): Music Waitlist Group: Participants in this group will serve as a control and will not receive any intervention until the study is completed. They will complete a baseline survey and a follow-up survey at four weeks. Some videos will be sent to this group after the study is completed, without tracking their usage.

INTERVENTIONS:
Behavioral: MIndfulness Listening to Jazz — All groups will complete a baseline and 4-week follow-up survey.
  Participants in Jazz Group 1 and Jazz Group 2 will engage in daily listening 4-week intervention.It is up to them if they want to listen to the daily recordings.
  Arms: MIndfullness and Jazz
Behavioral: Listening to Jazz — All groups will complete a baseline and 4-week follow-up survey.
  Participants in Jazz Group 1 and Jazz Group 2 will engage in daily listening 4-week intervention.They will have access to electronic audio recordings, with the order of listening labeled for each day. The recordings will increase gradually throughout the study, starting with about 10 minutes each day in the first week and reaching 30 minutes each day in the final week. The schedule is as follows: Week 1= 10 minutes, Week 2= 15 minutes, Week 3= 20 minutes Week 4= 30 minutes. It is up to them if they want to listen to the daily recordings.
  Arms: Jazz Only

SUMMARY:
Chronic pain, including spinal pain and osteoarthritis, is the leading cause of years lived with disability world-wide and the costliest health condition in the U.S. today. Compounding these concerns, opioid analgesics remain the primary pharmacological treatment for chronic pain. An estimated 21-29% of chronic pain patients receiving long-term opioid therapy develop opioid misuse, and opioid misuse portends addiction and overdose. Clearly, chronic pain patients need better, non-addictive treatment options designed to reverse the downward spiral of chronic pain.

DETAILED DESCRIPTION:
Group Assignments

Participants will be randomized into one of three groups.

1. Jazz Group 1: Participants in this group will watch an introduction to jazz appreciation video prior to the 4-week intervention.
2. Jazz Group 2 (Mindful Jazz) Group: Participants in this group will watch a video on mindful listening to jazz.
3. Music Waitlist Group: Participants in this group will serve as a control and will not receive any intervention until the study is completed. They will complete a baseline survey and a follow-up survey at four weeks. Some videos will be sent to this group after the study is completed, without tracking their usage.

Intervention

All groups will complete a baseline and 4-week follow-up survey.

Participants in Jazz Group 1 and Jazz Group 2 will engage in daily listening 4-week intervention.They will have access to electronic audio recordings, with the order of listening labeled for each day. It is up to them if they want to listen to the daily recordings.

ELIGIBILITY:
Inclusion Criteria:

1. Are 18+
2. Live in the US
3. Are an English-proficient adult with a chronic pain diagnosis (no restrictions placed on type)
4. Have a pain rating of four or greater in average pain on a 0-10 numeric rating scale in the preceding week
5. Have had pain for at least 3 months and for at least 15 days in the preceding 30 days
6. Have moderate to severe anxiety based on GAD-7

Exclusion Criteria:

1. Are currently using or have used prescription opioids in the past 3 months to minimize a known treatment confound and increase sample homogeneity
2. Have a current cancer diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity portion of The Pain, Enjoyment of Life and General Activity (PEG) scale | 4 weeks
  The Pain, Enjoyment of Life and General Activity (PEG) scale will be used to assess the magnitude of pain sensations experienced by participants in the past week. Range 0-10, where higher score equals more pain.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California Irvine, Irvine, California, United States